CLINICAL TRIAL: NCT01553708
Title: The Clinical Efficacy of Epidermal Growth Factor With Silver Sulfadiazine Cream Compared With Silver Zinc Sulfadiazine Cream on Acceleration of Partial Thickness Burn Wound Healing
Brief Title: Effect of EGF With Silver Sulfadiazine Cream Compared With Silver Zinc Sulfadiazine Cream for Treatment of Burn Wound
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: National Science and Technology Development Agency, Thailand (Other Government)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU0155
Record Dates: First submitted 2012-02-28; First posted 2012-03-14 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Deep Partial Thickness Burn
Keywords: Wound healing; Epithelialization; Safety
MeSH Terms: interventions — Epidermal Growth Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidermal growth factor with silver sulfadiazine cream (Experimental): Epidermal growth factor with silver sulfadiazine cream was applied to the experimental wounds completely and then covered with sterile gauze. The wound was cleaned every 24 h and the cream was then applied again after cleaning process.
  Interventions: Drug: Epidermal growth factor with silver sulfadiazine cream
- Silver zinc sulfadiazine cream (Active Comparator): Silver sulfadiazine cream was applied to cover the controlled-wound completely and then covered with sterile gauze. The wound was cleaned every 24 h and the cream was then applied again after cleaning process.
  Interventions: Drug: Silver zinc sulfadiazine cream

INTERVENTIONS:
Drug: Epidermal growth factor with silver sulfadiazine cream — Compare the duration for complete partial thickness burn wound healing between sample (epidermal growth factor with silver sulfadiazine cream) and control (silver zinc sulfadiazine cream)
  Arms: Epidermal growth factor with silver sulfadiazine cream
Drug: Silver zinc sulfadiazine cream — Compare the duration for complete partial thickness burn wound healing between sample (epidermal growth factor with silver sulfadiazine cream) and control (silver zinc sulfadiazine cream)
  Arms: Silver zinc sulfadiazine cream

SUMMARY:
Partial thickness burn wounds are most likely to heal within 2-3 weeks mainly by mechanism of epithelialization. However, it depends on the depth of the wounds and patient condition. Infection is one of the most common complications causing delay in wound healing which might affect to quality of patient's life. Generally, the standard treatment of partial thickness burn wound is topical 1% silver sulfadiazine cream. Previous studies had been reported the broad spectrum antimicrobial activity of silver sulfadiazine cream but it did not demonstrate the accelerating effect of wound healing. Therefore, the combination of substance which can promote wound healing to topical silver sulfadiazine cream might benefit for partial thickness burn wound treatment.

The objective of this study was to compare the results of partial thickness burn wound treatment at burn unit, Siriraj hospital with topical cream containing 1% silver sulfadiazine plus 6% epidermal growth factor (EGF) and 1% silver zinc sulfadiazine. The demographic data (age, sex, %body surface area burn), time of wound closure, pain and itching, dose and type of pain and itching medication, adverse effect of topical medication, some laboratory results and cost of expenses.

This is the prospective, double blinded, randomize-controlled study. The sample sizes were partial thickness burn wound patients who were treated at burn unit, Siriraj hospital. Patients were allocated into 2 groups receiving treatment with either topical silver sulfadiazine plus EGF or silver zinc sulfadiazine. All parameter data were analyzed with repeated measure ANOVA and independent t-test.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years.
* Partial thickness burn wound more than 20%TBSA.
* No underlying diseases that interfere wound healing such as chronic kidney disease, diabetes mellitus, liver disease, immunocompromised deficiency.
* In case of reproductive age woman, they have to control the birth rate at least 4 weeks before study.
* Patients who are willing to participate in the trial and to sign the informed consent form.

Exclusion Criteria:

* Immunocompromised defects
* Known allergy or hypersensitivity reaction to epidermal growth factor, silver sulfadiazine or other substances in formulation.
* Pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Pharm.D., Ph.D., Principal Investigator — Faculty of Pharmaceutical Sciences, Chulalongkorn University
Locations (1):
- Burn Unit, Siriraj Hospital, Bangkok, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited between December 2011 to May 2012 at Burn Unit, Siriraj Hospital, Bangkok, Thailand.
Pre-assignment Details: The subjects were excluded if inclusion criteria was not met or the other treatment was assigned by the physician.
Period: Overall Study
Arm/Group | Epidermal Growth Factor With Silver Sulfadiazine Cream | Silver Zinc Sulfadiazine Cream
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidermal Growth Factor With Silver Sulfadiazine Cream | Silver Zinc Sulfadiazine Cream | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.12 (13.72) | 37.71 (7.91) | 37.41 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  Thailand | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Time of Healing by Monitoring Duration (Days) at the Beginning of Treatment and the Day of Completely Epithelialization (Complete Epithelialization Means no Open Wound Exists as Confirmed by Two Surgeons).
Description: Time (days)for complete epithelialization (no open wound exists as determined by 2 surgeons) is the duration between the day of admission and the wound completely close without fluid leakage and are able to expose to environment without pain.
Time Frame: On 28th day after admission
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Epidermal Growth Factor With Silver Sulfadiazine Cream: Wounds treated with the cream containing epidermal growth factor and silver sulfadiazine evenly and covered with sterile gauze. Wounds were also cleaned with sterile normal saline daily and the cream was applied again after cleaning.
- Silver Zinc Sulfadiazine Cream: Wounds treated with the cream containing silver sulfadiazine evenly and covered with sterile gauze. Wounds were also cleaned with sterile normal saline daily and the cream was applied again after cleaning.
Arm/Group | Epidermal Growth Factor With Silver Sulfadiazine Cream | Silver Zinc Sulfadiazine Cream
Number analyzed (Participants) | 17 | 17
Days | 23.06 (5.21) [19 to 28] | 30.94 (7.34) [23 to 38]

2. Secondary Outcome: Clinical Safety of Epidermal Growth Factor With Silver Sulfadiazine Cream for Treatment of Partial Thickness Burn Wound.
Description: 1. Pain and itching assessment is evaluated by patients themselves in every time of wound observations using Visual Analog Scale.
  2. % Wound contraction.
  3. Time and type of analgesic or itching medication after treatment.
  4. Laboratory measurement such as CBC, blood glucose, electrolyte, hepatic and renal functions will be analyzed to find any changes or any systemic effect after treatment.
  5. Adverse reaction such as swelling, edema and redness at wound site.
Time Frame: On 28th day after admission
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Epidermal Growth Factor With Silver Sulfadiazine Cream | Silver Zinc Sulfadiazine Cream
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed and all samples have 18-60 years of age, this data cannot be applied for pediatrics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No